## **Study title**: Kupewa: Optimizing Implementation Strategies for Cervical Cancer Prevention

NCT number: NCT07015957

**Document date**: 2 July 2025

| | The conse | nt form sho | uld be signed only |
|---------------|------------|-----------------------|--------------------|
| | between_ | a) | rd |
| PROVIDER SURV | VEY CONSEN | BY NHSRC MIT (ENGLISH | ONLY) |

**Informed Consent: Provider Surveys** 

Research Study Title: Kupewa: Optimizing Strategies to Implement Provider Recommendation of HPV Vaccination for Adolescent Girls and Young Women with HIV in Malawi

This research study is a collaboration between investigators at New York University (U.S., Corrina Moucheraud), University of California Los Angeles (U.S., Risa Hoffman), and Partners in Hope (Malawi, Sam Phiri).

Introduction: You have been asked to participate in this study called "Kupewa: Optimizing Strategies to Implement Provider Recommendation of HPV Vaccination for Adolescent Girls and Young Women with HIV in Malawi" because you are a clinical officer, nurse, or medical assistant at this facility who interacts with parents or caregivers of girls aged 9-24 years. Your participation is entirely voluntary. You will now read more information about the study and are free to ask questions about anything you do not understand before deciding whether or not to participate.

**Purpose:** This study aims increase HPV vaccination in Malawi by increasing health workers' knowledge, skills, and memory to recommend HPV vaccination to girls and young women.

**Procedure:** If you consent and agree to take part, you will self-administer a baseline survey. The surveys will ask questions about knowledge and skills around talking with parents and young women about HPV vaccination. We will also ask your sex/gender, your cadre, and how long you've been in this role. You will repeat a similar survey two additional times during the study period; these surveys will repeat many of the same questions from the baseline survey plus your impressions of participating in the intervention. The information you provide will be connected across these three surveys for data analysis. In addition, we may contact you one year after the intervention ends for an additional post-intervention survey.

Hospitals and health centers that participate in this study will participate in an intervention that includes one or some combination of: 1) trainings for health workers, 2) coaching for health workers, or 3) a reminder system for health workers. Prior to beginning the study, each health facility was randomly assigned to one or more of these interventions. You will not know which of these interventions this health facility is participating in.

Participation in each of the three intervention-period surveys will take about 20 minutes (60 minutes total). You will be given MK18,000 for your time on all the surveys, MK6,000 for each survey. You must complete each survey in order to receive the associated payment, although you may skip any survey questions that you wish. There will be no costs for participating in the study or in the surveys.

**Benefits**: If you choose to participate in the research, your knowledge and skills to talk about HPV vaccination with your clients may be strengthened, which could have potential benefits to society. The knowledge gained from this study could potentially have a positive effect on health systems, particularly for regions that have a high burden of cervical cancer, like Malawi.



**Risks:** We do not anticipate any risks from participating in this research; if you do not want to answer any survey questions, you are free to skip them. No one can hear your responses since you will self-administer the survey. If you do not want to answer any question, you may skip it and will not be penalized for doing so.

Privacy and Confidentiality: The information you provide will be kept confidential. We will collect your name, your date of birth, and your phone number(s) (to contact you for the follow-up surveys), but if you do not want to answer any of these questions, you may skip it and will not be penalized for doing so. We will maintain the confidentiality and privacy of your data. Authorized representatives of the Malawi National Health Sciences Research Committee (NHSRC), the New York University (U.S.) Institutional Review Board, and others who are responsible for ensuring the rules related to research are followed, may need to review records of study participants. When the results of the research are published or discussed in meetings, no information will be included that would reveal your identity. Any data related to the study will be kept on an encrypted computer in a locked cabinet in a locked office at Partners in Hope or NYU. Your personal data will only be retained as long as reasonably necessary for this research. Afterwards, PIH will either delete your personal data or anonymize your data to ensure you are no longer identifiable. These de-identified data may be kept for use in future research, and may be shared with the research community to advance scholarly knowledge. We plan to deposit the de-identified data in the Qualitative Data Repository, which is an online database that helps researchers share the information that they learn from their studies with one another, so we can all keep learning together. All information that could identify you will be removed before sharing the data or using it for other research studies. We will not ask you for additional permission before sharing the information.

Participation and Withdrawal: Your participation in the research is voluntary. You may stop at any time or chose to not answer any of the questions. Additionally, the research investigator may stop your participation in the discussion, if he or she feels this is best for you.

**Study Approval:** Institutional review boards that have oversight in this research include the National Health Sciences Research Committee in Lilongwe, Malawi, and the NYU Institutional Review Board, New York, USA (contacts below).

In the event of a research-related problem, please contact the investigators (contact information below). If you have any questions about the research, please feel free to contact either of the individuals listed below.

Pericles Kalande

Research Coordinator, Partners in Hope Clinic Area 36 Plot 8 M1 Road South Lilongwe, Malawi <u>pkalande@pihmalawi.com</u>

Telephone: 0994424889

Corrina Moucheraud, ScD, MPH

New York University, School of Global Public Health, Department of Public Health Policy and Management

c.moucheraud@nyu.edu

Telephone: +1-212-992-6129

2

| | | | | | BETWEEN HELESTICATION OF THE REST. TABLE TO A SEC. |
|---|---|---|---|---|---|
| | This consent | form | should be | signed | enty 1 |
| between and | | | | | |
| | Approved by | NHSR | C. Malaw | ion | |

If you have questions about your rights as a research subject or if you wish to voice any problems or concerns you may have about the study to someone other than the researchers, please contact:

Dr. Evelyn Chitsa Banda
The National Health Sciences Research Committee in Lilongwe, Malawi
P.O. Box 30377
Lilongwe 3, Malawi.
Telephone 0999-936-937

If you have questions about your rights as a research participant or if you believe you have been harmed from the research, please contact the NYU Human Research Protection Program at +1-212-998-4808 or ask.humansubjects@nyu.edu

I have read (or someone has read to me) the information provided above. I have been given an opportunity to ask questions and all of my questions have been answered to my satisfaction. I have been given a copy of this form.

BY CHECKING THE BOX BELOW, I WILLINGLY AGREE TO PARTICIPATE IN THE RESEARCH:

☐ I have read this information and consent to participate in this research as described.